CLINICAL TRIAL: NCT02787473
Title: A Phase II Study of Pemetrexed Plus Cisplatin With Concurrent Radiation Therapy Followed by Every-21-Day Docetaxel Consolidation in Patients With Inoperable Stage IIIA/B Squamous Cell Lung Cancer
Brief Title: A Study of Pemetrexed Plus Cisplatin With Concurrent Radiation Therapy Followed by Docetaxel Consolidation in Patients With Inoperable Squamous Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HZCH-2016-10
Record Dates: First submitted 2016-04-22; First posted 2016-06-01 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Squamous Cell Lung Cancer
Keywords: Squamous cell lung cancer; Pemetrexed; Radiosensitivity
MeSH Terms: interventions — Pemetrexed; Cisplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- pemetrexed+carboplatin/cisplatin+radiation therapy->docetaxel (Experimental): Patients received pemetrexed 500mg/m2 days 1,29+cisplatin 25 mg/m2 days 1-3,29-31 + Radiation 6000 cGy (200 cGy/day). Patients with complete response(CR), partial response(PR) or stable disease(SD) with manageable toxicity received docetaxel 60 mg/m2 days 57,78.
  Interventions: Drug: pemetrexed; Drug: cisplatin; Radiation: thoracic radiation therapy; Drug: docetaxel

INTERVENTIONS:
Drug: pemetrexed — Pemetrexed 500mg/m2 IV on day 1 every 4 weeks for 2 cycles
Drug: cisplatin — Cisplatin 25mg/m2 IV on day 1-3 every 4 weeks for 2 cycles
  Other Names: platinol
Radiation: thoracic radiation therapy — Chemoradiotherapy, radiation 60Gy with 2 cycles of pemetrexed+ carboplatin/cisplatin
Drug: docetaxel — Docetaxel 60 mg/m2 IV on day 57 every 3 weeks for 2 cycles
  Other Names: taxotere

SUMMARY:
To evaluate the efficacy and toxicity of patients with inoperable squamous cell lung cancer treated with pemetrexed plus cisplatin with concurrent radiation therapy followed by docetaxel consolidation. An exploratory biomarker analysis in blood and tumor samples is also planned.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed stage IIIA/ IIIB squamous cell lung cancer;
* All sites of disease must be amenable to definitive radiotherapy;
* Age 18 years to 75 years;
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2;
* Forced expiratory volume in 1 second(FEV1)> 0.75L;
* No previous chest radiotherapy, immunotherapy or biotherapy;
* Adequate bone marrow, liver and renal function, as specified below: Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L; Hemoglobin ≥ 8 g/dL; Platelets ≥ 100 x 109/L; Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN) ; Aspartate transaminase(AST) and alanine Transaminase(ALT) ≤ 2.5 x ULN or ≤ 5 x ULN if liver metastases are present; Serum creatinine ≤ 1.5 x upper limit of normal or creatinine clearance ≥ 60ml/min for patients with creatinine levels above institutional normal.
* For women of child-bearing potential, negative pregnancy test within 14 days prior to starting treatment
* Men and women of childbearing age must be willing to use effective contraception while on treatment and for at least 3 months thereafter;
* Patients and their family signed the informed consents;

Exclusion Criteria:

* Active infection;
* History of significant cardiac disease (unstable angina, congestive heart failure, myocardial infarction within the previous 6 months, ventricular arrhythmias);
* Malnutrition (loss of ≥ 20% of the original body weight);
* Performance status: 3-4;
* Sensor or motor neuropathy > grade I;
* Second primary malignancy, except for non-melanoma skin cancer;
* Psychiatric illness or social situation that would preclude study compliance;
* Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2016-10; Primary Completion 2019-10 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | 3 years

SECONDARY OUTCOMES:
Overall Survival | 3 years
Local control rate | 3 years
The short-term quality of life (QOL) assessed using FACT-E score | 4 months
  FACT-E score at the 4 months after docetaxel consolidation therapy
Rate of CTCAE grade 2 or higher radiation pneumonitis | 1 years
  The investigators will assess the rate of symptomatic radiation pneumonitis in patients who received the radiation therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China